CLINICAL TRIAL: NCT06604208
Title: Double-blind, Randomized, Placebo-controlled Trial to Explore the Improvement of Sleep Quality of Insomnia Patients with "Binaural Beats"
Brief Title: Improvement of Sleep Quality of Insomnia Patients with "Binaural Beats"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202401052B0
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-08

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Binaural Beats (Experimental)
  Interventions: Device: Binaural Beats
- Placebo (Sham Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Binaural Beats — The binaural beat device is a health product that is not classified as a medical device. It functions similarly to a music box, providing different frequencies through physiological and psychological induction. This process offers binaural beat information to the Reticular Activating System (RAS) for potential changes in consciousness. The binaural beat frequencies are designed to match the brainwave frequency of light sleep, specifically 3.4 Hz (θ waves), with a base frequency of 440 Hz. The device uses three types of background music-piano music, light music, and string music-as experimental materials.
  The binaural beat device offers three modes, allowing users to select different modes based on their comfort and listening preferences. This study requires that the binaural beats be listened to for at least 30 minutes. The device has a built-in app for continuous playback, so users can connect the power and listen throughout the night.
  Arms: Binaural Beats
Device: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if binaural beat works to treat chronic insomnia in adults. It will also learn about the safety of binaural beat. The main questions it aims to answer are:

What medical problems do participants have when using binaural beat? Researchers will compare binaural beat to a placebo to see if binaural beat works to treat chronic insomnia.

Participants will:

Using binaural beat or a placebo every day for 2 weeks Keep a diary and actigraphy of their insomnia symptoms Visit the clinic after 2 weeks testing for checkups and tests

DETAILED DESCRIPTION:
As the pace of society accelerates, people are under increasing mental stress, which can lead to emotional instability and even insomnia. Insomnia is a common sleep disorder characterized by difficulty falling asleep, poor sleep quality, and early awakening. Studies have shown that chronic insomnia is closely related to diseases such as hypertension and type 2 diabetes and can lead to impaired daytime functioning and mood disorders. The prevalence of insomnia is high, affecting about 10% of the global population. In Taiwan, the prevalence of chronic insomnia is 11.3%, with higher rates observed in women and the elderly. However, many insomnia patients receive only medication, despite the potential side effects of long-term use of sleeping pills. Therefore, exploring the effectiveness of non-pharmacological treatments for insomnia is crucial. In recent years, various non-invasive and non-pharmacological therapies such as mindfulness therapy, acupressure therapy, and acupuncture therapy have gained attention. Overall, the demand for research and treatment of insomnia is increasing.

Additionally, some emerging therapies such as Schumann wave therapy and binaural beat therapy are being explored in research. The former has been shown to improve sleep quality, while the latter has shown potential for enhancing sleep. Binaural beats play a significant role in sleep medicine. This auditory stimulation involves hearing slightly different frequencies in each ear, influencing the brain through the brainstem and reticular activating system to create a new frequency, thereby improving sleep quality. Research indicates that dynamic binaural beats (DBB) can effectively shorten sleep latency and reduce heart rate variability, helping to enhance sleep quality. Furthermore, the application of binaural beats has expanded to the field of insomnia treatment, aiming to help insomnia patients improve sleep quality and increase safety. These research findings suggest that binaural beats may be a non-invasive, effective, non-pharmacological treatment option for sleep support.

The binaural beat device is a health product that is not classified as a medical device. It functions similar to a music box, providing different frequencies through physiological and psychological induction. This process offers binaural beat information to the Reticular Activating System (RAS) for potential changes in consciousness. The binaural beat frequencies are designed to match the brainwave frequency of light sleep, specifically 3.4 Hz (θ waves), with a base frequency of 440 Hz. The device uses three types of background music-piano music, light music, and string music-as experimental materials.

The binaural beat device offers three modes, allowing users to select different modes based on their comfort and listening preferences. This study requires that the binaural beats are listened to for at least 30 minutes. The device has a built-in app for continuous playback, so users can connect the power and listen throughout the night.

ELIGIBILITY:
Inclusion Criteria:

* Gender: No restrictions, Age: Between 20 and 75 years.
* Meets the criteria for insomnia as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5):

  1. Difficulty sleeping and insomnia occurring at least 3 nights per week.
  2. Insomnia and sleep difficulties persisting for at least 3 months.
* The participant has signed the informed consent form.

Exclusion Criteria:

* Individuals who are unable to complete the consent form, undergo testing, and attend regular follow-up visits as required by the study.
* Individuals with severe physical illnesses or post-surgical conditions, such as heart disease or metabolic disorders.
* Individuals with severe psychiatric disorders, including schizophrenia, major depressive disorder, severe anxiety disorder, bipolar disorder, dementia, or substance use disorders; or severe neurological conditions, such as stroke or epilepsy.
* Individuals with other severe sleep disorders, such as severe sleep apnea.
* Individuals who are unable to maintain a stable medication dosage during the trial period, particularly with ongoing treatments.
* Patients deemed unsuitable for participation in the trial by the principal investigator.
* Patients who are unable to adhere to sleep hygiene practices or who cannot refrain from using electronic devices before bedtime.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | baseline, week3, week 7
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized questionnaire designed to assess sleep quality and patterns over a one-month period. The PSQI has a scoring range from 0 to 21, with higher scores indicating worse sleep quality. The questionnaire is divided into seven components, each addressing different aspects of sleep, such as sleep duration, disturbances, and daytime dysfunction. The sum of these component scores gives the overall PSQI score.
Actigraphy | baseline, week1-2
  Actigraphy is a non-invasive method used to monitor and assess sleep patterns and circadian rhythms. It involves wearing a small, wristwatch-like device called an actigraph, which measures movement over extended periods, typically one week or longer. By analyzing the data collected, researchers or clinicians can estimate sleep duration, sleep onset, wake times, and periods of restlessness. Actigraphy is particularly useful for studying sleep in naturalistic settings, providing an objective measure of sleep-wake cycles without requiring the individual to stay in a sleep lab. It is often used to assess sleep disorders, such as insomnia or circadian rhythm disturbances, and can be an essential tool for both clinical evaluations and sleep research.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | baseline, week3, week 7
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire used to assess an individual's general level of daytime sleepiness. The ESS asks respondents to rate their likelihood of falling asleep in eight different situations that are commonly encountered in daily life. The scale ranges from 0 to 24, with higher scores indicating greater levels of daytime sleepiness. Higher scores on the ESS reflect a worse outcome in terms of sleep health.
Beck Depression Inventory (BDI) | baseline, week3, week 7
  The Beck Depression Inventory (BDI) is a widely used self-report questionnaire designed to assess the severity of depressive symptoms in individuals. The BDI consists of 21 items, each corresponding to a specific symptom of depression, such as sadness, pessimism, or loss of interest. Respondents rate each item on a scale from 0 to 3, resulting in a total score that ranges from 0 to 63. Higher scores on the BDI indicate more severe depressive symptoms, with specific thresholds used to categorize the severity of depression (e.g., minimal, mild, moderate, or severe). Therefore, higher scores represent a worse outcome, signaling more intense depression.
Beck Anxiety Inventory (BAI) | baseline, week3, week 7
  The Beck Anxiety Inventory (BAI) is a self-report questionnaire used to assess the severity of anxiety symptoms in individuals. The BAI consists of 21 items, each describing a common symptom of anxiety, such as nervousness, dizziness, or fear of losing control. Respondents rate how much they have been bothered by each symptom over the past week on a scale from 0 to 3. The total score ranges from 0 to 63, with higher scores indicating more severe anxiety. Specific score ranges help categorize the level of anxiety (e.g., minimal, mild, moderate, or severe), making higher scores reflective of a worse outcome in terms of anxiety severity.
Short Form (36) Health Survey (SF-36) | baseline, week3, week 7
  The Short Form (36) Health Survey (SF-36) is a widely used questionnaire designed to assess overall health-related quality of life across multiple dimensions. It includes 36 items that measure eight key health concepts: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health perceptions. The SF-36 generates scores for each of these domains, as well as two summary measures: physical and mental health. Scores for each domain and summary measure range from 0 to 100, with higher scores indicating better health and quality of life. Therefore, higher scores on the SF-36 represent a better outcome.
Sleep diary | baseline, week1-3, week 7
  A Sleep Diary is a self-reported tool used to track sleep patterns and behaviors over a period of time, typically one to two weeks. It includes daily entries where individuals record various aspects of their sleep, such as bedtime, wake time, sleep onset latency, number and duration of awakenings, and overall sleep quality. The data collected is used to identify sleep patterns, irregularities, and potential sleep disorders, making it a valuable resource for both clinical assessments and personal sleep management.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Shu Huang, MD, PhD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal SD, Landon BE. Patterns in Outpatient Benzodiazepine Prescribing in the United States. JAMA Netw Open. 2019 Jan 4;2(1):e187399. doi: 10.1001/jamanetworkopen.2018.7399. PMID 30681713
- [Background] Belisheva NK, Popov AN, Petukhova NV, Pavlova LP, Osipov KS, Tkachenko SE, Varanova TI. [Qualitative and quantitative assessment of exposure to geomagnetic field variations on the functional status of the human brain]. Biofizika. 1995 Sep-Oct;40(5):1005-12. Russian. PMID 8555283
- [Background] Buscemi N, Vandermeer B, Friesen C, Bialy L, Tubman M, Ospina M, Klassen TP, Witmans M. The efficacy and safety of drug treatments for chronic insomnia in adults: a meta-analysis of RCTs. J Gen Intern Med. 2007 Sep;22(9):1335-50. doi: 10.1007/s11606-007-0251-z. Epub 2007 Jul 10. PMID 17619935
- [Background] Colzato LS, Barone H, Sellaro R, Hommel B. More attentional focusing through binaural beats: evidence from the global-local task. Psychol Res. 2017 Jan;81(1):271-277. doi: 10.1007/s00426-015-0727-0. Epub 2015 Nov 26. PMID 26612201
- [Background] Galvez G, Recuero M, Canuet L, Del-Pozo F. Short-Term Effects of Binaural Beats on EEG Power, Functional Connectivity, Cognition, Gait and Anxiety in Parkinson's Disease. Int J Neural Syst. 2018 Jun;28(5):1750055. doi: 10.1142/S0129065717500551. Epub 2017 Nov 13. PMID 29297265
- [Background] Wahbeh H, Calabrese C, Zwickey H. Binaural beat technology in humans: a pilot study to assess psychologic and physiologic effects. J Altern Complement Med. 2007 Jan-Feb;13(1):25-32. doi: 10.1089/acm.2006.6196. PMID 17309374
- [Background] Zampi DD. Efficacy of Theta Binaural Beats for the Treatment of Chronic Pain. Altern Ther Health Med. 2016 Jan-Feb;22(1):32-8. PMID 26773319